CLINICAL TRIAL: NCT03385538
Title: Clopidogrel Response and CYP2C19 Genotype in Ischemic Stroke Patients
Acronym: CLOGIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-003548-38
Record Dates: First submitted 2017-08-21; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clopidogrel non-responders (Experimental): Increasing doses og Clopidogrel depending on PRU values measured on VerifyNow
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — increasing doses of clopidogrel depending on PRU values (75-300 mg)

SUMMARY:
Personalized therapy as prophylaxis in ischemic stroke patients is not yet an option. From patients with ischemic heart disease, we know that patients with in vitro high on treatment platelet reactivity (HTPR) have an increased risk of stent thrombosis following per-cutaneous coronary intervention. Other studies have shown association of CYP2C19 genotypes with different responses to the anti platelet drug Clopidogrel. We measure HTPR in ischemic stroke patients on increasing doses of clopidogrel and investigate the CYP2C19 genotype for each patient.

DETAILED DESCRIPTION:
Background: Clopidogrel (CLO) is a pro-drug metabolized in the liver by the Cytochrom-P450 system to its active component. Studies in acute ischemic stroke (IS) patients have proven that genetic differences in coding of an enzyme responsible for the metabolism of CLO (CYP2C19) results in different response to CLO when tested in the blood. An American study in cardiac patients have shown an association between the genotype and the CLO-response to different dosages of CLO, meaning that patients who are non-responders to low dosages of CLO may be responders to higher CLO dosages. Furthermore, the study showed that patients with a distinct genotype does not gain CLO response even at high CLO dosages (300 mg/day).

Perspective: The study will have an impact on the patient, the relatives and the social economy. The project answers if it is possible to give personalized therapy to IS patients securing the best possible prophylactic treatment for each single patient. Hereby reducing the risk of early death, disability and dependency. The project determines the genetic distribution of CYP2C19 alleles in the Danish IS population and determine the association between genotype and CLO-response in clinically relevant dosages in a Caucasian population of IS patients.

Objective: To determine the correlation between genotype and Clopidogrel response to different CLO dosage and to determine the distribution of different alleles of CYP2C19 genotypes in a Danish IS population.

Hypothesis: CLO response is determined by CYP2C19 genotype, and there is a correlation between drug-response and CYP2C19 genotype.

Method: Systematic recording of data on 103 IS patients receiving prophylactic treatment with CLO 75 mg/day.

Genotype is determined in collaboration with Division of Clinical Biochemistry, Dept. of Diagnostics, Glostrup Hospital determining the CYP2C19 genotype *1(wild-type), *2(Loss Of Function=LOF) and *17(Gain Of Function=GOF). CLO responder status is determined using the VerifyNow P2Y12 assays.

Patients receiving CLO 75 mg/day who are non-responders when testing with VerifyNow P2Y12 assays have a blood sample for genetic testing. Patients carrying the *2 genotype on one or both alleles are CLO responder status tested on increasing doses of CLO, rising 75 mg/day every 14 days (150/225/300 mg) until maximum CLO 300 mg/day. Responder status is tested at the end of every second week, before increasing dosage. If the patient is CLO responder on the tested dose (150/225/300 mg) or non-responder on CLO 300 mg/day, the patient is ended in the study and switched to treatment with ASA in combination with Dipyramidole.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke diagnosis
* treatment with clopidogrel 75 mg/day

Exclusion Criteria:

* increased risk of bleeding
* treatment with NOAC, vitamin K antagonist or other antiplatelet drug than clopidogrel
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who has clopidogrel HTPR | 7 days
  Clopidogrel responder status measured with VerifyNow
Number of patients who are carriers of CYP2C19 loss-of-function alleles | 1 day
  Genotyping patients for different loss-of-function CYP2C19 alleeles (*2, *3)
Number of patients who are carriers of P2Y12-receptor loss-of-function alleles | 1 day
  genotyping patients for different loss-of-function P2Y12 receptor alleeles

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Rath, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, dept of neurology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No